CLINICAL TRIAL: NCT05778994
Title: Use of the Intorus Device as a Therapeutic Tool for the Control of Anxiety Before the Exams in Occupational Therapy Students of the University of Extremadura
Brief Title: Use of Intorus to Control Anxiety Before Exams in Students at the University of Extremadura
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Extremadura (Other)
Responsible Party: Principal Investigator, Blanca González Sanchez, DOCTOR. PRINCIPAL INVESTIGATOR, University of Extremadura
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2023.ALUMNOS.INTORUS
Record Dates: First submitted 2023-01-30; First posted 2023-03-22 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: STUDENT; Anxiety Disorders
Keywords: STUDENTS; ANXIETY; OCCUPATIONAL THERAPY
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXPERIMENTAL (Experimental): Group that performs therapy with intorus
  Interventions: Device: INTORUS
- CONTROL (No Intervention): Group without intervention

INTERVENTIONS:
Device: INTORUS — Exercise protocol with intorus
  Arms: EXPERIMENTAL

SUMMARY:
The goal of this clinical trial is to assess the possible efficacy of the INTORUS device as an element to reduce test anxiety in university students. The main question[s] it aims to answer are:

Can the INTORUS device be used as a tool to reduce anxiety? Once informed, those participants who meet the inclusion/exclusion criteria and sign the informed consent to participate in the study will be randomly divided into two groups. The randomization procedure will be carried out using the OxMaR (Oxford Minimization and Randomization) software.

All participants will be given the Sociodemographic Questionnaire, Self-efficacy Scale and anxiety questionnaire prior to the start of the study.

DETAILED DESCRIPTION:
The population is made up of students of the Degree in Occupational Therapy during the 2nd semester of the 2022-2023 academic year.

The initial sample size will be approximately 70 participants.

- Process

Once informed, those participants who meet the inclusion/exclusion criteria and sign the informed consent to participate in the study will be randomly divided into two groups. The randomization procedure will be carried out using the Oxford Minimization and Randomization software.

All participants will be given the Sociodemographic Questionnaire, Self-efficacy Scale and anxiety questionnaire prior to the start of the study.

The participants of the experimental group will carry out a weekly exercise session with INTORUS aimed at reducing anxiety in the period between March 1, 2023 and May 10, 2023.

On the day of the final exam for the subject, all students will repeat the anxiety measurement questionnaire and the perceived self-efficacy scale minutes before the final exam for the subject.

Once the intervention period is over, a questionnaire will be passed to the professionals participating in the study to assess the usefulness of the device, the degree of satisfaction with it and the usefulness of the therapies applied.

ELIGIBILITY:
Inclusion Criteria:

* Students of the Degree in Occupational Therapy at the University of Extremadura.
* Students who are going to study the Degree in Occupational Therapy in person.

Exclusion Criteria:

* Not meeting the inclusion criteria
* Not wanting to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Changes in the BECK anxiety questionnaire over 3 months | Measures before starting the intervention. through study completion, an average of 3 months.
  Questionnaire to measure anxiety. The questionnaire consists of 21 questions, providing a range of scores between 0 and 63. The suggested cut-off points for interpreting the result obtained are as follows:
  00-21 - Very low anxiety 22-35 - Moderate anxiety over 36 - Severe anxiety

SECONDARY OUTCOMES:
Changes in the Perceived self-efficacy scale in academic situations | Measures before starting the intervention. through study completion, an average of 3 months.
  Scale to measure participants' perceived self-efficacy in academic situations. the scale is structured with 10 items, wherein factorial loads are higher than .63 (with the exception of item 9); with high reliability α = .91 and temporal stability (10 weeks) r = .91. higher scores mean a worse outcome.
Changes in the questionnaire for the assessment of anxiety before exams | Measures before starting the intervention. through study completion, an average of 3 months.
  Questionnaire to measure participants' level of test anxiety. a standardized measurement scale for test anxiety, consists of 20 items that separate worry and emotionality and, at the same time, yields total score of examination anxiety. higher scores mean a worse outcome.

OTHER OUTCOMES:
Participant satisfaction questionnaire | Through study completion, an average of 3 months
  Questionnaire to measure patient satisfaction with the protocol. higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Blanca González Sáchez, Doctor, Principal Investigator — Universidad de Extremadura
Locations (1):
- Blanca Gonzalez Sanchez, Cáceres, Spain

IPD SHARING:
Plan to Share IPD: No